CLINICAL TRIAL: NCT00293072
Title: Pilot Study of Rituximab Therapy for Systemic Lupus Erythematosus (SLE) and Vasculitis Resistant to Conventional Therapy
Brief Title: Pilot Study of Rituximab Therapy for Systemic Lupus Erythematosus (SLE) and Vasculitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Roche Pharma AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pilot study of Rituximab
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2006-02-17 (Estimated); Status verified 2005-10

CONDITIONS: Systemic Lupus Erythematosus; ANCA Associated Vasculitis
Keywords: Rituximab, ANCA, vasculitis, lupus,
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
Lupus and vasculitis are autoimmune conditions which can be life threatening. In order to treat these conditions toxic therapies such as cyclophosphamide and steroids are often required. These standard treatments are associated with significant side effects. Furthermore a proportion of patient do not respond to these conventional therapies. Newer safer therapies are being sought. Rituximab is a drug that eliminates B cell from the blood. B cells are one part of the human immune system that helps prevent infections. Abnormal activity of the immune system is responsible for autoimmune disease although the exact mechanisms in lupus and vasculitis are not yet established. Rituximab is liscenced as a treatment for a form of B cell cancer called non-Hodgkins Lymphoma and has a good safety track record when used in this context. It has recently been used to treat some autoimmune conditions with positive results. In this pilot study we wish to assess the effectiveness and safety of rituximab in patients with lupus and vascultis that are resistant to conventional therpies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SLE or ANCA associated vasculitis
2. Active disease refractory to 6 months conventional therapy with cyclophosphamide, prednisolone and at least one other immunosupressive agent ( or a lesser period if this therapy cannot be tolerated)
3. Age 18-70

Exclusion Criteria:

1. HbeAg or HCV Ab positive or known HIV positivity ( HIV testing not necessary for this study)
2. Pregnancy, inadequate contraception or lactation
3. Malignancy
4. Current enrolment in pother clinicla trials -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-03; Study Completion 2005-05

PRIMARY OUTCOMES:
1. Clinical remission at 6 or 12 months
2. Absence of a severe life threatening adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Ken Smith, Principal Investigator — Cambridge Institute for Medical Research, Addenbrooke's Hospital; David Jayne, Principal Investigator — Lupus and Vasculitis Service, Addenbrooke's Hospital
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom